CLINICAL TRIAL: NCT03206021
Title: Phase I/Ib Trial of COmbined 5'aZacitidine and Carboplatin for Recurrent/Refractory Pediatric Brain and Solid Tumors
Brief Title: COZMOS:Phase I/Ib Trial of Combined 5'Azacitidine and Carboplatin for Recurrent/Refractory Pediatric Brain/Solid Tumors
Acronym: COZMOS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Vijay Ramaswamy, Staff Physician, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OZM-077
Record Dates: First submitted 2017-06-21; First posted 2017-07-02 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Childhood CNS Tumor; Ependymoma, Recurrent Childhood; Childhood Solid Tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Ependymoma | interventions — Azacitidine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I Dose-escalation (Experimental): 5'azacytidine will be administered on Days 1-7 at a dose of 75mg/m2/day, followed by escalating doses of Carboplatin on Day 14 in a rolling 6 design. Carboplatin will be dosed initially at AUC 4. Dose level -1 will reduce 5'azacytidine to 50mg/m2/day.
  Interventions: Drug: 5 Azacytidine
- Posterior Fossa Ependymoma Expansion Arm (Experimental): 5'azacytidine will be administered on days 1-7 and carboplatin will be administered on day 14 at the maximum tolerated dose achieved in the Phase I dose escalation to 20 patients with recurrent/refractory posterior fossa ependymoma.
  Interventions: Drug: 5 Azacytidine
- Recurrent Brain and Solid Tumour Expansion Arm (Experimental): 5'azacytidine will be administered on days 1-7 and carboplatin will be administered on day 14 at the maximum tolerated dose achieved in the Phase I dose escalation up to 12 patients with recurrent/refractory brain and solid tumour.
  Interventions: Drug: 5 Azacytidine

INTERVENTIONS:
Drug: 5 Azacytidine — Dose escalation of carboplatin combined with 5'azacytidine
  Other Names: Carboplatin

SUMMARY:
Many pediatric brain and solid tumors have altered epigenetic landscapes, and altered DNA methylation. As such this study is a Phase I/Ib study of combined 5'Azacitidine with an escalating dose of carboplatin for all recurrent/refractory pediatric brain and solid tumors. The phase I component will establish with maximum tolerated dose of carboplatin with azacytidine. An expansion cohort will be recruited of up to 30 patients will follow consisting of 20 recurrent posterior fossa ependymoma and 10 recurrent supratentorial ependymoma.

DETAILED DESCRIPTION:
Aberrant DNA methylation is frequently observed in many pediatric solid tumors, but in particularly several entities such as ependymoma, medulloblastoma, embryonal tumor with multilayered rosettes, atypical/teratoid rhabdoid tumor, neuroblastoma and wilm's tumor have promoter hypermethylation. Treatment with DNMTi (DNA methyltransferase inhibitors) agents such as 5-azacytidine has been shown to be safe and efficacious in adult myelodysplastic syndromes, causing significant decreased DNA methylation in blood, with maximum effect at day 15 of each cycle. However, monotherapy with DNMTi has been shown to result in resistance in leukamia's and efficacy in solid tumours is limited. Synergy between DNMTi and platinum agents has shown promise in pre-clinical models including pediatric ependymoma, and in addition, the combination of demethylating agents with carboplatin has provided promising results in platinum resistant ovarian cancers. However, this approach has not been applied to pediatric solid malignancies, which are attractive targets due to their frequent epigenetic dysregulation.

Platinums are the backbone of therapy for most pediatric solid tumors, and as such it is an attractive hypothesis that part of the reason for resistance to upfront therapies is platinum resistance. Specifically, ependymoma's are highly chemoresistant tumors and studies in preclinical models of ependymoma support that this chemoresistance can be overcome with DNMTi.

There is a clear medical need for new therapies, particularly for relapsed solid tumors, specifically brain tumors. Although pre-clinical data from our group and others suggests DNA demethylase inhibitors to be promising therapies for high risk ependymoma, medulloblastoma and ETMR (embryonal tumor with multilayered rosettes), 5'azacitidine monotherapy has been disappointing in clinical studies of adult solid tumours. Previous studies have suggested that platinum therapy can be effectively combined with azacitidine therapy and based on adult studies, maximum demethylation occurs approximately 5-10 days after treatment with 5'azacitidine. As such combination of azacitidine and carboplatin is a rationale therapy for several pediatric brain tumours, particularly those with a hypermethylated phenotype.

Two phases of the study will be conducted. The Phase I will establish the maximum tolerated dose of carboplatin and 5'azacytidine in a rolling 6 design. 5'azacytidine will be administered on Days 1-7 followed by Carboplatin on Day 15. The initial dose level will be 5'Azacytidine 75mg/m2/day for 7 days with Carboplatin administered on Day 15 at AUC (Area under curve) 4. Carboplatin will be dose escalated to a maximum of AUC 6, or de-escalated to AUC 3. The Phase Ib will be an ependymoma specific expansion cohort at the established MTD (maximum tolerated dose), to determine the feasibility and initial efficacy of the combination of carboplatin and 5'azacytidine in patients with recurrent/refractory posterior fossa and supratentorial ependymoma.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than the age of 1 year and under age 18 at the time of study enrolment
2. Recurrent or refractory brain or solid tumor, including recurrent or refractory ependymoma
3. Tissue from diagnosis or resection prior to registration must be available (either flash frozen tissue or an FFPE block)
4. Previous therapy with carboplatin will be permitted
5. Failed first line treatment (surgery, radiation therapy or chemotherapy) and should not be eligible for treatment with curative potential.
6. Be at least 4 weeks from the completion of myelosuppressive chemotherapy and/or biologic agents before starting day 1 of this study treatment
7. Be at least 14 days from the completion of radiation therapy and MIBG before starting day 1 of this study treatment
8. Be at least 3 months post hematopoetic stem cell rescue following myeloablative therapy before starting day 1 of this study treatment
9. Must have visible disease on imaging. Resection of visible disease is permitted while on study after two cycles including achievement of a gross total resection. If a resection is performed while on study, fresh frozen tissue should be submitted for analysis.
10. Concurrent medications will be limited to supportive medications/agents including but not limited to anti-emetics, steroids, analgesics and non-enzyme inducing anticonvulsants. Strong inducers of the P450 system will not be permitted. Other concurrent medications require approval of the study Sponsor.
11. Ability of the parent and/or child to understand and the willingness to sign a written informed consent document
12. Karnofsky ≥ 50 for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age (See Appendix I for the Karnofsky-Lansky Scores). Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score. Patients with posterior fossa syndrome/cerebellar mutism demonstrating clear improvement post-surgically can be enrolled based on physician discretion
13. Adequate hepatic, renal, marrow and cardiac function as defined below within 28 days prior to cycle 1 day 1:

    * Serum creatinine within normal institutional limits or creatinine clearance greater than 60mL/min
    * Serum bilirubin <1.5 times upper limit of institutional normal. Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis
    * AST, ALT and Alkaline Phosphatase <3 times upper limit of institutional normal. If liver metastases are present, then <5 times upper limit of normal is permitted.
    * Normal QTc interval at screening ECG (baseline echocardiogram is not required)
    * Adequate marrow function defined below within 14 days prior to cycle 1 day 1:

      * Leukocytes greater than or equal to 1000 x106/L
      * Absolute neutrophil count greater than or equal to 0.75 x109/L
      * Platelets greater than or equal to 75 x109/L
      * Hemoglobin greater than or equal to 10g/dL (may be transfused).

Exclusion Criteria:

1. Female patient who is pregnant or breast feeding (Lactating females must agree not to breast feed while taking azacitidine) or with childbearing potential and not willing to use a double method of contraception up to 3 months after the end of study treatment. Male patient who is not willing to use a barrier method of contraception up to 6 months after the end of study treatment.
2. Patients may not be receiving any other investigational agents within 30 days prior to day 1 of protocol treatment
3. Prior therapy with a DNA demethylase inhibitor
4. Evidence of cardiac toxicity (shortening fraction below 28%; shortening fraction measures and ratios the change in the diameter of the left ventricle between the contracted and relaxed states)
5. Abnormal coagulation parameters (PT >15 seconds, PTT>40 seconds, and/or INR >1.5)
6. Significant active cardiac disease within the previous 6 months including:

   * NYHA class 3 or 4 CHF
   * Unstable angina
   * Myocardial infarction
7. Known or suspected hypersensitivity to azacitidine or mannitol carboplatin
8. Previous carboplatin exposure is not an exclusion criteria but previous allergic reaction to carboplatin will exclude enrolment.
9. Patient must not require use of enzyme inducing anticonvulsants; patients who are receiving an enzyme inducing anticonvulsant must be able to switch to a non-enzyme inducing anticonvulsant such as Levetiracetam, Clobazam, Lacosamide, Valproate or Topiramate at least 2 weeks prior to study enrolment.
10. Uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
11. Active viral infection with HIV or hepatitis type B or C Patients with advanced malignant hepatic tumors
12. Patients with advanced malignant hepatic tumors

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Establish maximum tolerated dose of carboplatin in combination with 5'azacytidine | 1 year
  Number of participants with treatment-related adverse events as assessed by the CTCAE4.0

SECONDARY OUTCOMES:
Characterization of the pharmacodynamics of 5'-azacitidine in combination with carboplatin | 3 years
  Plasma pharmacodynamics will be assessed using methylation profiling of whole blood collected before and after administration of 5'Azacytidine, and after administration of carboplatin.
Assessment of intratumoral DNA demethylation as a preliminary indication of biological efficacy of this combination. | 3 years
  Where feasible, two cycles of 5'azacytidine and carboplatin will be administered prior to a biopsy and/or gross total resection, and intratumoral DNA methylation profiles will be generated to determine the degree of intratumoral DNA demethylation.
Assessment of disease response as a preliminary indication of efficacy of this combination against recurrent, refractory pediatric brain and solid tumors | 3 years
  Response to therapy, particularly in ependymoma will be evaluated to determine if a larger Phase II study is warranted.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Ramaswamy, MD PhD FRCPC, Principal Investigator — The Hospital for Sick Children; Peter Dirks, MD PhD FRCSC, Principal Investigator — The Hospital for Sick Children; Eric Bouffet, MD, Principal Investigator — The Hospital for Sick Children; Daniel Morgenstern, MD PhD, Principal Investigator — The Hospital for Sick Children
Locations (17):
- Children's National Medical Center, Washington D.C., District of Columbia, United States
- Australia (8):
  - Royal Children's Hospital Melbourne, Melbourne, Victoria
  - Women's and Children's Hospital, Adelaide
  - Monash Children's Hospital, Clayton
  - John Hunter Children's Hospital, Lambton
  - Perth Children's Hospital, Perth
  - Queensland Children's Hospital, South Brisbane
  - Sydney Children's Hospital, Sydney
  - Children's Hospital at Westmead, Westmead
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre hospitalier universitaire Sainte-Justine, Montreal, PQ
  - Montreal Children's Hospital, Montreal, PQ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mack SC, Witt H, Piro RM, Gu L, Zuyderduyn S, Stutz AM, Wang X, Gallo M, Garzia L, Zayne K, Zhang X, Ramaswamy V, Jager N, Jones DT, Sill M, Pugh TJ, Ryzhova M, Wani KM, Shih DJ, Head R, Remke M, Bailey SD, Zichner T, Faria CC, Barszczyk M, Stark S, Seker-Cin H, Hutter S, Johann P, Bender S, Hovestadt V, Tzaridis T, Dubuc AM, Northcott PA, Peacock J, Bertrand KC, Agnihotri S, Cavalli FM, Clarke I, Nethery-Brokx K, Creasy CL, Verma SK, Koster J, Wu X, Yao Y, Milde T, Sin-Chan P, Zuccaro J, Lau L, Pereira S, Castelo-Branco P, Hirst M, Marra MA, Roberts SS, Fults D, Massimi L, Cho YJ, Van Meter T, Grajkowska W, Lach B, Kulozik AE, von Deimling A, Witt O, Scherer SW, Fan X, Muraszko KM, Kool M, Pomeroy SL, Gupta N, Phillips J, Huang A, Tabori U, Hawkins C, Malkin D, Kongkham PN, Weiss WA, Jabado N, Rutka JT, Bouffet E, Korbel JO, Lupien M, Aldape KD, Bader GD, Eils R, Lichter P, Dirks PB, Pfister SM, Korshunov A, Taylor MD. Epigenomic alterations define lethal CIMP-positive ependymomas of infancy. Nature. 2014 Feb 27;506(7489):445-50. doi: 10.1038/nature13108. Epub 2014 Feb 19. PMID 24553142
- [Result] Ramaswamy V, Hielscher T, Mack SC, Lassaletta A, Lin T, Pajtler KW, Jones DT, Luu B, Cavalli FM, Aldape K, Remke M, Mynarek M, Rutkowski S, Gururangan S, McLendon RE, Lipp ES, Dunham C, Hukin J, Eisenstat DD, Fulton D, van Landeghem FK, Santi M, van Veelen ML, Van Meir EG, Osuka S, Fan X, Muraszko KM, Tirapelli DP, Oba-Shinjo SM, Marie SK, Carlotti CG, Lee JY, Rao AA, Giannini C, Faria CC, Nunes S, Mora J, Hamilton RL, Hauser P, Jabado N, Petrecca K, Jung S, Massimi L, Zollo M, Cinalli G, Bognar L, Klekner A, Hortobagyi T, Leary S, Ermoian RP, Olson JM, Leonard JR, Gardner C, Grajkowska WA, Chambless LB, Cain J, Eberhart CG, Ahsan S, Massimino M, Giangaspero F, Buttarelli FR, Packer RJ, Emery L, Yong WH, Soto H, Liau LM, Everson R, Grossbach A, Shalaby T, Grotzer M, Karajannis MA, Zagzag D, Wheeler H, von Hoff K, Alonso MM, Tunon T, Schuller U, Zitterbart K, Sterba J, Chan JA, Guzman M, Elbabaa SK, Colman H, Dhall G, Fisher PG, Fouladi M, Gajjar A, Goldman S, Hwang E, Kool M, Ladha H, Vera-Bolanos E, Wani K, Lieberman F, Mikkelsen T, Omuro AM, Pollack IF, Prados M, Robins HI, Soffietti R, Wu J, Metellus P, Tabori U, Bartels U, Bouffet E, Hawkins CE, Rutka JT, Dirks P, Pfister SM, Merchant TE, Gilbert MR, Armstrong TS, Korshunov A, Ellison DW, Taylor MD. Therapeutic Impact of Cytoreductive Surgery and Irradiation of Posterior Fossa Ependymoma in the Molecular Era: A Retrospective Multicohort Analysis. J Clin Oncol. 2016 Jul 20;34(21):2468-77. doi: 10.1200/JCO.2015.65.7825. Epub 2016 Jun 6. PMID 27269943